CLINICAL TRIAL: NCT03987750
Title: A Phase 3, Double-blind, Placebo-controlled, Parallel-group Study to Assess the Efficacy and Safety of 2 Doses of Safinamide Compared to Placebo in the Treatment of LID in PD Patients With Motor Fluctuations
Brief Title: Safinamide for Levodopa-induced Dyskinesia (PD-LID)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: drug development plan has been updated
Sponsor: Zambon SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Z7219L04
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2019-06

CONDITIONS: Dyskinesia, Drug-Induced; Parkinson Disease
MeSH Terms: conditions — Dyskinesia, Drug-Induced; Parkinson Disease | interventions — safinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Safinamide 100mg (Experimental): Participants randomized to the 100 mg study arm will receive 100 mg safinamide methanesulfonate film-coated tablets once daily during Week 1 (2 x 50 mg active tablets plus 1 placebo tablet) and throughout the rest of the study safinamide
  Interventions: Drug: Safinamide Methanesulfonate 100mg
- Safinamide 150mg (Experimental): Participants randomized to the 150 mg study arm will receive 100 mg methanesulfonate film-coated tablets once daily during Weeks 1 and 2 (2 x 50 mg active tablets plus 1 placebo tablet), and 150 mg methanesulfonate film-coated tablets once daily(3 x 50 mg active tablets) from Week 3 and throughout the rest of the study
  Interventions: Drug: Safinamide Methanesulfonate 150mg
- Placebo (Placebo Comparator): Participants randomized to the placebo arm will receive Safinamide Methanesulfonate matching placebo film-coated tablets once daily (3 x placebo tablets)
  Interventions: Drug: Safinamide Methanesulfonate matching placebo

INTERVENTIONS:
Drug: Safinamide Methanesulfonate 150mg — 150 mg (free base)
  Arms: Safinamide 150mg
Drug: Safinamide Methanesulfonate 100mg — 100 mg (free base)
  Arms: Safinamide 100mg
Drug: Safinamide Methanesulfonate matching placebo — placebo
  Arms: Placebo

SUMMARY:
This will be a prospective, multi-center, randomized, double-blind, parallel group, placebo-controlled study, in participants with PD who are on a stable regimen of dopaminergic medication and have at least mild levodopa-induced dyskinesia. Eligible participants will be randomized to one of three treatment groups to receive adjunctive daily treatment with either safinamide 100 mg, safinamide 150 mg or placebo in a 1:1:1 ratio. Outcome will be assessed after 26 weeks of treatment.

DETAILED DESCRIPTION:
Trial participation will be up to a maximum duration of 32 weeks and will comprise:

* Screening period (up to 4 weeks) for screening assessments;
* Two weeks titration period: participants randomized to the 100 mg study arm will receive 100 mg during Week 1 and throughout the rest of the study; participants randomized to the 150 mg study arm will receive 100 mg during Weeks 1 and 2 , and 150 mg from Week 3 and throughout the rest of the study; participants randomized to the placebo arm will receive identical placebo tablets.
* Twenty-four weeks maintenance period during which patients receive their randomized treatment as an adjunct to their standard anti-PD medications, which should remain unaltered. End of treatment evaluations will be performed at the end of Week 26 or at early discontinuation
* A telephone follow-up call will be performed 2 weeks after the end of treatment to assess adverse events and concomitant medications

ELIGIBILITY:
Inclusion Criteria:

1. Male and female participants aged 30 years and above at the time of signing the informed consent;
2. Female participants may participate if they are not of child bearing potential (post-menopausal with no periods for at least one year, or surgically sterilized);
3. Women of child bearing potential (WOCBP) may participate if they are not pregnant, not breastfeeding, and agree to follow the contraceptive guidance during the treatment period and for at least 30 days after the last dose of study intervention;
4. A diagnosis of Parkinson's disease consistent with the UK PD Brain Bank Society and MDS Clinical Diagnostic Criteria;
5. Levodopa immediate release and/or controlled release, given at least 3 times daily, on a stable regimen for at least 4 weeks prior to screening;
6. Participants may also be taking benserazide, catcechol O methyl transferease (COMT) inhibitors and dopamine agonists, the dose of which must be stable for at least 4 weeks prior to screening;
7. Predictable peak dose dyskinesia of at least mild severity and causing at least mild disability as defined as a score of ≥2 on the MDS UPDRS questions 4.1 and 4.2 at screening and at least two 30 minute periods of ON time with troublesome dyskinesia recorded in 24 hour PD home diaries performed in each of the two days prior to the randomization visit;
8. Participants with motor fluctuations with at least three 30 minute periods in OFF (for a total of 1.5 hours per waking day) in each of the two consecutive 24 hour home diaries completed at the end of the screening period in the 48 hours prior to Day 1
9. Provided written informed consent as described in Appendix 1 which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol, prior to the study screening procedures commencing.

Exclusion Criteria:

1. Participants with secondary or atypical parkinsonian syndrome
2. Participants with solely diphasic dyskinesia without peak dose dyskinesia
3. History of neurosurgical procedure for Parkinson's disease, including stereotactic surgery and Deep Brain Stimulation (DBS).
4. Treatment with monoamine oxidase inhibitors, amantadine pethidine, dextromethorphan, fluoxetine, fluvoxamine in the 8 weeks prior to the screening visit
5. Concomitant use of selective serotonin reuptake inhibitors (SSRIs), serotonin norepinephrine reuptake inhibitors (SNRIs), tricyclic/tetracyclic antidepressants may be permitted but used at the lowest doses.
6. Participants who are unable to complete the home diary and have 2 consecutive 24-hour periods with more than 4 missing periods per 24 hours in the diary, completed at the end of the screening period, in the 48 hours prior to Day 1
7. History of major psychiatric disease eg bipolar disorder, severe depression, schizophrenia or other psychosis.
8. Current history of Impulse Control Disorder
9. History of drug and/or alcohol abuse within 12 months prior to screening (DSM-V criteria)
10. History of dementia (DSM-V criteria) or cognitive impairment MMSE < 24 at screening
11. Ophthalmologic history of the following conditions: albinism, uveitis, retinitis pigmentosa, retinal degeneration, active retinopathy, severe progressive diabetic retinopathy, inherited retinopathy or family history of hereditary retinal disease.
12. Moderate or severe hepatic impairment with transaminases >2 times upper limit of normal (ULN) or bilirubin 1.5 times ULN
13. Any clinically significant or unstable medical or surgical condition that, in the opinion of the investigator, might preclude safe completion of the study or might affect the results of the study.
14. Use of any investigational drug within 30 days prior to screening or 5 half-lives, whichever is the longest.
15. Allergy/sensitivity or contraindications to the investigational medicinal product (IMP) or their excipients.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-10 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Assess the effect of two doses of safinamide on reducing levodopa-induced dyskinesia | 26 weeks
  Change from Baseline to Week 26 in levodopa-induced dyskinesia based on UDysRS total score. The UDysRS is a dyskinesia rating scale from 0-104; it evaluates involuntary movements associated with PD. A higher score indicates more severe PD

SECONDARY OUTCOMES:
Assess the effect of two doses of safinamide on ON time with No Dyskinesia | 26 weeks
  Change from Baseline (Day 1 prior to start of study intervention) to Week 26 total daily ON time with No dyskinesia based on PD Home Diary. A PD home diary is used to score 5 different conditions : ASLEEP, OFF, ON (ie, had adequate control of PD symptoms) without dyskinesia, ON with non-troublesome dyskinesia, and ON with troublesome dyskinesia.
Assess the effect of two doses of safinamide on ON time with non-troublesome dyskinesia | 26 weeks
  Change from Baseline (48 hours prior to Day 1) to Week 26 based on PD Home Diary in total daily ON time with non-troublesome dyskinesia. A PD home diary is used to score 5 different conditions : ASLEEP, OFF, ON (ie, had adequate control of PD symptoms) without dyskinesia, ON with non-troublesome dyskinesia, and ON with troublesome dyskinesia.
Assess the effect of two doses of safinamide on ON time with troublesome dyskinesia | 26 weeks
  Change from Baseline (48 hours prior to Day 1) to Week 26 based on PD Home Diary in total daily ON time with troublesome dyskinesia. A PD home diary is used to score 5 different conditions : ASLEEP, OFF, ON (ie, had adequate control of PD symptoms) without dyskinesia, ON with non-troublesome dyskinesia, and ON with troublesome dyskinesia.
To assess the effect of two doses of safinamide on ON time with any dyskinesia (troublesome or non-troublesome) | 26 weeks
  Change from Baseline (48 hours prior to Day 1) to Week 26 based on PD Home Diary in total daily ON time with any dyskinesia (troublesome or non-troublesome). A PD home diary is used to score 5 different conditions : ASLEEP, OFF, ON (ie, had adequate control of PD symptoms) without dyskinesia, ON with non-troublesome dyskinesia, and ON with troublesome dyskinesia.
To assess the effect of two doses of safinamide on sleep time | 26 weeks
  Change from Baseline (48 hours prior to Day 1) to Week 26 based on PD Home Diary in total daily sleep time. A PD home diary is used to score 5 different conditions : ASLEEP, OFF, ON (ie, had adequate control of PD symptoms) without dyskinesia, ON with non-troublesome dyskinesia, and ON with troublesome dyskinesia.
To assess the effect of two doses of safinamide on Movement Disorder Society-Sponsored Unified Parkinson's Disease Rating Scale (MDS-UPDRS) total score and sub-scores | 26 weeks
  Change from Baseline (Day 1 prior to start of study intervention) to Week 26 in MDS-UPDRS total score and sub-scores. The MDS-UPDRS is divided into 4 parts. In each part, all items are rated on a scale from 0 (normal) to 4 (severe impairment); Part I assesses 15 items of non-motor aspects of experiences of daily living; Part II comprises 13 items evaluating the impact of PD on patients' activities of daily living (ADL) over the week prior to the visit such as speech, salivation, swallowing, eating, handwriting, dressing, turning in bed, walking; part III assesses the motor abilities in PD patients at the time of the visit; Part IV assesses motor complications of therapy, such as dyskinesias, motor fluctuations.
To assess the effect of two doses of safinamide on Clinician Global Impression of Change (CGIc) | 26 weeks
  Clinician Global Impression of Change (CGIc) at Week 26. CGI-C is a 7-point scale used by Investigator to rate patient's overall improvement using a range of responses from 1 (very much improved) through to 7 (very much worse).
To assess the effect of two doses of safinamide on Patient Global Impression of Change (PGIc) | 26 weeks
  Patient Global Impression of Change (CGIc) at Week 26. PGI-C is a 7-point scale depicting a patient's rating of overall improvement using a range of responses from 1 (very much improved) to 7 (very much worse).
To assess the effect of two doses of safinamide on PDQ-39 summary index | 26 weeks
  Change from Baseline (Day 1 prior to start of study intervention) to Week 26 in PDQ-39 summary index. The PDQ-39 is a specific tool to assess quality of life in PD. Comprises 39 items divided into eight dimensions: mobility, activities of daily living (ADLs), emotional well-being, stigma, social support, cognition, communication and physical discomfort, where scores range from 0-100, with the higher, the worse the perception of quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Keywood, MD, Study Director — Zambon SpA